CLINICAL TRIAL: NCT03634358
Title: Bipolar Scissors Versus Classic Method for Circumcision
Brief Title: Bipolar Scissors for Circumcision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, yousef ahmed el-ayman, assistant lecturer of general surgery, MD Candidate, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZagazigUH
Record Dates: First submitted 2018-01-13; First posted 2018-08-16 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Male Circumcision
Keywords: bipolar; scalpel; foreskin; prepuce

STUDY DESIGN:
Intervention Model Description: Comparing Outcomes of two different surgical techniques between two groups
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bipolar scissors group (Active Comparator): Group of male infants undergoing circumcision using bipolar scissors to separate the foreskin
  Interventions: Procedure: Bipolar scissors
- Classic scalpel group (Active Comparator): Group of male infants undergoing circumcision using classic scalpel to separate the foreskin, and sutures to control bleeding
  Interventions: Procedure: classic scalpel

INTERVENTIONS:
Procedure: Bipolar scissors
  Arms: Bipolar scissors group
Procedure: classic scalpel
  Arms: Classic scalpel group

SUMMARY:
comparing the outcomes of using bipolar scissors for male circumcision to the classic scalpel method

DETAILED DESCRIPTION:
A prospective, randomized study, comparing two different techniques for pediatric male circumcision: the bipolar diathermy scissors technique with that of a classic scalpel technique. Study included male infants from 40 days old up to 18 month old. They were reviewed regarding Operative time, bleeding, complications, postoperative pain and morbidity. Differences in the outcome were compared.

ELIGIBILITY:
Inclusion Criteria:

* Male infant between 40 days and 18 month old
* parents' request and approval of circumcision

Exclusion Criteria:

* previous attempts of circumcision or revision cases
* bleeding tendency
* congenital anomalies involving genitalia
* age below 40 days (expected Vit. K deficiency) or above 18 month old.

Ages: 40 Days to 18 Months | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-01-10 (Actual); Study Completion 2018-01-10 (Actual)

PRIMARY OUTCOMES:
Post-operative bleeding | A week
  occurrence of active bleeding after circumcision

SECONDARY OUTCOMES:
Post-operative pain | A week
  pain after operation as assessed and described by parents (through a questionnaire) by the Neonatal/Infant Pain Scale (NIPS): It is composed of six (6) indicators.
  * facial expression
  * cry
  * breathing patterns
  * arms
  * legs
  * state of arousal Each behavioral indicator is scored with 0 or 1 except "cry", which has three possible descriptors therefore, being scored with a 0, 1 or 2. Infants should be observed for one minute in order to fully assess each indicator. Total pain scores range from 0-7. Pain Level is determined as: 0-2 = mild to no pain. 3-4 = mild to moderate pain >4 = severe pain
wound complications | Two weeks
  occurrence of infection, necrosis or skin loss around wound
Cosmetic outcome | Two month
  Presence or absence of scar
Operative time | Operative time
  Duration of procedure of both techniques
Over or under correction | 2 month
  Excessive or insufficient removal of foreskin (presence of redundant skin or compression of penile length)

REFERENCES:
- [Background] Mendez-Gallart R, Estevez E, Bautista A, Rodriguez P, Taboada P, Armas AL, Pradillos JM, Varela R. Bipolar scissors circumcision is a safe, fast, and bloodless procedure in children. J Pediatr Surg. 2009 Oct;44(10):2048-53. doi: 10.1016/j.jpedsurg.2009.06.008. PMID 19853772